CLINICAL TRIAL: NCT05520723
Title: Multicenter, Open-label, Single Arm, Phase II Clinical Trial to Improve Sacituzumab Govitecan's Tolerance in Patients With Metastatic Triple-Negative or Luminal Breast Cancer.
Brief Title: Preventive stRategy for IMMU132-relatED AEs in TNBC or Luminal Breast Cancer- PRIMED
Acronym: PRIMED
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedSIR (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEDOPP445; 2022-001397-61 (EudraCT Number)
Record Dates: First submitted 2022-07-19; First posted 2022-08-30 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Triple Negative Breast Cancer; Breast Cancer; Advanced HR+/HER2- Breast Cancer
Keywords: Advanced TNBC; Sacituzumab govitecan; Tolerance; Prophylaxis; Advanced HR+/HER2-
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms | interventions — sacituzumab govitecan; Loperamide; Granulocyte Colony-Stimulating Factor; Filgrastim

STUDY DESIGN:
Masking Description: Open label, single-arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sacituzumab Govitecan + Loperamide + G-CSF (Experimental): Upon meeting all selection criteria, patients enrolled in the study will receive the combination of:
  Sacituzumab govitecan :10 mg/kg, intravenously (IV) on Days 1 and 8 every 21-day cycle .
  This treatment will continue until disease progression, unacceptable toxicity, or physician's/patient's decision.
  Loperamide : 2 mg orally (PO), twice a day (BID), or 4 mg once a day (QD) during three consecutive days after administration of sacituzumab govitecan, (D2, D3, D4 and D9, D10, D11) during the first two cycles (consider extending to the next cycle at the discretion of the physician).
  G-CSF : 30 MU subcutaneously (SC) QD during two consecutive days, 48 hours after administration of sacituzumab govitecan (D3, D4 and D10, D11) during the first two cycles (consider extending to the next cycle at the discretion of the physician).
  Interventions: Drug: Sacituzumab govitecan; Drug: Loperamide; Drug: Granulocyte Colony-Stimulating Factor

INTERVENTIONS:
Drug: Sacituzumab govitecan — Upon meeting all selection criteria, patients enrolled in the single-arm study will receive the combination of: sacituzumab govitecan and prophylaxis (loperamide and G-CSF).
  Sacituzumab govitecan :10 mg/kg, intravenously (IV) on Days 1 and 8 every 21-day cycle . This treatment will continue until disease progression, unacceptable toxicity, or physician's/patient's decision.
  Other Names: Trodelvy
Drug: Loperamide — Loperamide : 2 mg orally (PO), twice a day (BID), or 4 mg once a day (QD) during three consecutive days after administration of sacituzumab govitecan, (D2, D3, D4 and D9, D10, D11) during the first two cycles (consider extending to the next cycle at the discretion of the physician).
  Other Names: Imodium
Drug: Granulocyte Colony-Stimulating Factor — G-CSF : 30 MU subcutaneously (SC) QD during two consecutive days, 48 hours after administration of sacituzumab govitecan (D3, D4 and D10, D11) during the first two cycles (consider extending to the next cycle at the discretion of the physician).
  Other Names: Filgrastim; Neupogen

SUMMARY:
This is a multicenter, open-label, single-arm, multicohort, two-stage optimal Simon's design, phase II clinical trial that is designed to improve the tolerance of sacituzumab govitecan in patients with unresectable locally advanced or metastatic triple negative breast cancer (TNBC) or Luminal breast cancer, refractory to at least one, and no more than two, prior standard of care chemotherapy regimens in this setting that is not amenable to resection with curative intent.

The goal of this study is to evaluate the safety of sacituzumab govitecan in combination with loperamide and G-CSF in pretreated patients with unresectable locally advanced or metastatic TNBC or Luminal breast cancer.

DETAILED DESCRIPTION:
The hypothesis of this study is that the prophylactic administration of loperamide (for diarrhea) and G-CSF therapies (for neutropenia) would avoid these undesirable effects when patients are treated with sacituzumab govitecan, thus decreasing the rate of dose reduction or discontinuation, and significantly improving patients' quality of life.

The main objectives of this study are:

Primary objective:

- To evaluate the incidence of diarrhea and neutropenia in patients with unresectable locally advanced or metastatic TNBC or Luminal breast cancer treated with sacituzumab govitecan in combination with loperamide and G-CSF.

Secondary objectives:

* To determine the safety and tolerability of the study regimen in this patient population.
* To determine the efficacy of the study regimen in this patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form (ICF) prior to participation in any study-related activities.
2. Patients aged ≥18 years at the time of signing ICF.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Life expectancy of ≥ 12 weeks.
5. Unresectable locally advanced or metastatic disease documented by computerized tomography (CT) scan or magnetic resonance imaging (MRI) that is not amenable to resection with curative intent.
6. All patients must have been previously treated with taxanes regardless of disease stage (adjuvant, neoadjuvant, or advanced), unless contraindicated for a given patient.
7. Refractory to at least one, and no more than two, prior standard of care chemotherapy regimens for unresectable locally advanced or MBC. Earlier adjuvant or neoadjuvant therapy for more limited disease will be considered as one of the required prior regimens if the development of unresectable locally advanced or metastatic disease occurred within a 12-month period after completion of chemotherapy or immunotherapy (e.g., adjuvant pembrolizumab).
8. For TNBC patient only:

   a.) Histologically confirmed TNBC per American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) criteria based on local testing on the most recent analyzed biopsy. Triple-negative is defined as <1% expression for estrogen receptor (ER) and progesterone receptor (PgR) and negative for human epidermal growth factor receptor 2 (HER2) (0-1+ by IHC or 2+ and negative by in situ hybridization [ISH) test].
9. For HR positive luminal breast cancer patients only:

   1. Confirmed diagnosis of estrogen receptor (ER)[+] and/or progesterone receptor (PR)[+] (with ≥1% positive stained cells according to National Comprehensive Cancer Network [NCCN] and American Society of Clinical Oncology [ASCO] guidelines) and human epidermal growth factor receptor 2 (HER2)- negative (0 or 1+ by immunohistochemistry [IHC] or 2+ and negative by in situ hybridization [ISH] test) breast cancer in the advanced setting.
   2. Refractory to at least 1 prior anticancer hormonal treatment and at least 1 CDKi4/6 in the metastatic setting.
10. Measurable or non-measurable, but evaluable disease, as per RECIST v.1.1. Patients with bone-only metastases are also eligible.
11. Brain MRI must be done for patients with suspicion of brain metastases and patient must have stable central nervous system (CNS) disease for at least 4 weeks after local therapy, without neurological symptoms, and off anticonvulsants and steroids for at least 2 weeks before first dose of study treatment.
12. Adequate hematologic counts without transfusional or growth factor support within 2 weeks before of study drug initiation (hemoglobin ≥ 9 g/dL, ANC ≥ 1500/mm3, and platelets ≥ 100,000/μL).
13. Adequate renal and hepatic function (creatinine clearance of ≥ 60 ml/min, may be calculated using Cockcroft-Gault equation; bilirubin ≤ 1.5 x ULN, AST and ALT ≤ 3.0 x ULN or 5 x ULN if known liver metastases).
14. Resolution of all acute AEs of prior anti-cancer therapy to grade 1 as determined by the NCI-CTCAE v.5.0 (except for alopecia or other toxicities not considered a safety risk for the patient at investigator discretion).
15. Male patients and female patients of childbearing potential who engage in heterosexual intercourse must agree to use institution specified method(s) of contraception.
16. Patients must have completed all prior cancer treatments at least 2 weeks* prior to randomization including chemotherapy (includes also endocrine treatment), radiotherapy, and major surgery.

    * Prior antibody treatment for cancer must have been completed at least 3 weeks prior to randomization.

Exclusion Criteria:

1. Prior treatment with topoisomerase 1 inhibitors as a free form or as other formulations.
2. Patients with carcinomatous meningitis or leptomeningeal disease.
3. Known hypersensitivity reaction to any investigational or therapeutic compound or their incorporated substances.
4. Patients with Gilbert's disease.
5. Patients known to be HIV positive, hepatitis B positive, or hepatitis C positive.
6. Participants with non-melanoma skin cancer or carcinoma in situ of the cervix are eligible, while participants with other prior malignancies must have had at least a 3-year disease-free interval.
7. Known history of unstable angina, myocardial infarction, or cardiac heart failure present within 6 months of study initiation or clinically significant cardiac arrhythmia (other than stable atrial fibrillation) requiring anti-arrhythmia therapy or history of QT interval prolongation.
8. Known history of clinically significant active Chronic obstructive pulmonary disease (COPD), or other moderate-to-severe chronic respiratory illness present within 6 months of study initiation.
9. Known history of clinically significant bleeding, intestinal obstruction, or gastrointestinal perforation within 6 months of study initiation.
10. Active or prior documented inflammatory bowel disease (i.e. Crohn's disease, ulcerative colitis, or a preexisting chronic condition resulting in baseline grade ≥1 diarrhea).
11. Infection requiring antibiotic use within 1 week of randomization.
12. Other concurrent medical or psychiatric conditions that, in the Investigator's opinion, may be likely to confound study interpretation or prevent completion of study procedures and follow-up examinations.
13. Women who are pregnant or lactating.
14. Concomitant participation in other interventional clinical trial. Note: Patients participating in observational studies are eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-02-06 (Actual); Primary Completion 2023-10-18 (Actual); Study Completion 2025-11-05 (Actual)

PRIMARY OUTCOMES:
Incidence of grade ≥2 diarrhea | Baseline up to end of 2nd cycle (day 42)
  The rate of patients with grade ≥ 2 diarrhea is defined as the number of patients with diarrhea grade 2 to 5 the first 2 cycles of treatment by the number of patients in the analysis set per 100.
  The adverse events will be assessed by the Investigator and with severity determined using defined and graded according CTCAE v.5.0. The adverse events without the severity grade reported will be considered as grade 3.
Incidence of grade ≥3 neutropenia | Baseline up to end of 2nd cycle (day 42)
  The rate of patients with grade ≥ 3 neutropenia is defined as the number of patients with neutropenia grade 3 to 5 the first 2 cycles of treatment by the number of patients in the analysis set per 100.
  The adverse events will be assessed by the Investigator and with severity determined using defined and graded according CTCAE v.5.0. The adverse events without the severity grade reported will be considered as grade 3.

SECONDARY OUTCOMES:
Incidence of all grades and grade ≥3 diarrhea. | Until EoS (26 months after study initiation)
  Adverse events during the study treatment will be coded according with Medical Dictionary for Regulatory Activities (MedDRA). NCI-CTCAE toxicity grades will be utilized for classifying severity. The adverse events without the severity grade reported will be considered as grade 3.
Incidence of all grades and grade ≥3 neutropenia. | Until EoS (26 months after study initiation)
  Adverse events during the study treatment will be coded according with Medical Dictionary for Regulatory Activities (MedDRA). NCI-CTCAE toxicity grades will be utilized for classifying severity. The adverse events without the severity grade reported will be considered as grade 3.
Incidence of febrile neutropenia and additional adverse events (AEs) as per NCI-CTCAE v.5.0. | Until EoS (26 months after study initiation)
  Adverse events during the study treatment will be coded according with Medical Dictionary for Regulatory Activities (MedDRA). NCI-CTCAE toxicity grades will be utilized for classifying severity. The adverse events without the severity grade reported will be considered as grade 3.
Discontinuation rate | Until EoS (26 months after study initiation)
  The discontinuation rate is defined as the proportion of participants discontinued to any cause relative to the number of patients in the analysis set. The reasons for study discontinuation and the period from the treatment initiation to the time of discontinuation will be also reported.
Dose reduction rate | Until EoS (26 months after study initiation)
  The dose reduction rate is defined as the proportion of participants with dose reduction relative to the number of patients in the analysis set. The reasons for dose reduction and the period from the treatment initiation to the time of the first dose reduction will be also reported.
Objective response rate (ORR) | Until EoS (26 months after study initiation)
  Objective response rate is defined as the proportion of participants with complete response or partial response relative to the number of patients in the analysis set. It will be also calculated only for patients with measurable disease at baseline. Participants who do not have on-study radiographic tumor re-evaluation, who received anti-tumor treatment other than the study medication, who died, progressed, or dropped out for any reason prior to reaching an objective response will be counted as non-responders in the assessment of ORR. Tumor response will be defined as best response based on local investigator's assessment according to RECIST v1.1.
Clinical benefit rate (CBR) | Until EoS (26 months after study initiation)
  Clinical benefit rate is defined as the proportion of participants with objective response, or stable disease ≥24 weeks relative to the number of patients in the analysis set. Non-complete response/non-progressive disease will be considered as stable disease. Clinical benefit will be also calculated only for patients with measurable disease at baseline. Participants who do not have on-study radiographic tumor re-evaluation, who received anti-tumor treatment other than the study medication, who died, progressed, or dropped out for any reason prior to reaching an objective response, or stable disease ≥24 weeks will be counted as without clinical benefit. Tumor response will be defined as best response based on local investigator's assessment according to RECIST v1.1 (Appendix 2).
Duration of response (DoR) | Until EoS (26 months after study initiation)
  Duration of response is defined as the time from the first documentation of objective tumor response to the first documentation of disease progression, death due to any cause or treatment discontinuation, whichever occurs first. Duration of response will be calculated in patients with objective response as [the date response ended (i.e., date of PD, death or discontinuation) - first objective response date +1)]/30.4.
Time to response (TtR) | Until EoS (26 months after study initiation)
  Time to response is defined as the period from the treatment initiation to time of the first objective tumor response (tumor shrinkage of ≥30%) observed for patients who achieved an objective response, as determined locally by the investigator through the use of RECIST v.1.1. The length of time to response will be calculated in patients with objective response as [(Objective response or censor date) - treatment initiation date +1]/30.4.
Best percentage of change from baseline in the size of target tumor lesions. | Until EoS (26 months after study initiation)
  Best percentage of change from baseline in the size of target tumor lesions, defined as the biggest decrease, or smallest increase if no decrease will be observed, as determined locally by the investigator using RECIST v.1.1. Participants who do not have on-study radiographic tumor re-evaluation, who received anti-tumor treatment other than the study medication, who died, progressed, or dropped out for any reason prior to reaching an objective response, or stable disease ≥24 weeks will be counted as not available. The analysis will be performed on patients with measurable disease at baseline.
Progression free survival (PFS) | Until EoS (26 months after study initiation)
  Progression-free survival is defined as the period from the date of treatment initiation to the date of the first documentation of objective progressive disease determined locally by investigator or death due to any cause in absence of documented progressive disease. Participants lacking an evaluation of tumor response after treatment initiation will have their progression-free survival time censored on the date of treatment initiation with the duration of a day. The length of progression-free survival will be calculated as [(progression, death date or censor date) - treatment initiation date +1]/30.4. Progression will be determined locally by the investigator using RECIST v.1.1. Objective PD is defined as 20% increase in the sum of diameters of target lesions above the smallest sum observed. The sum must also demonstrate and absolute increase of at least 5 mm or unequivocal progression of existing non-target lesions or the appearance of new lesion.

CONTACTS AND LOCATIONS:
Locations (10):
- Spain (10):
  - Hospital Universitario A Coruña, A Coruña, A Coruna
  - Hospital Universitario General de Catalunya, Sant Cugat del Vallès, Barcelona
  - Hospital Universitario Donostia, San Sebastián, Donostia
  - Hospital Arnau de Vilanova, Lleida, Lleida
  - Hospital Quiron San Camilo- Ruber Juan Bravo, Madrid, Madrid
  - Hospital Quirón Valencia, Valencia, Valencia
  - Hospital de Sant Joan Despí - Moises Broggi, Barcelona
  - Hospital Universitario Clínico San Cecilio de Granada, Granada
  - Hospital Ramón y Cajal, Madrid
  - Hospital Universitario Virgen del Rocio, Seville